CLINICAL TRIAL: NCT06252012
Title: The Effect of Cervical Cancer Awareness Education Based on Mobile Application on Women's Attitudes and Behaviors Regarding Cervical Cancer Prevention and Early Diagnosis
Brief Title: The Effect of Cervical Cancer Awareness Education Based on Mobile Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Principal Investigator, Fatma Nur Sena, Lecturer, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS-2305
Record Dates: First submitted 2023-05-04; First posted 2024-02-09 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Cervix Cancer; Cancer Awareness; Mobile Application; HPV; Nurse's Role
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: A mobile application developed to increase awareness of cervical cancer among 60 women in the intervention group who met the sample criteria was implemented.
Who Masked: Participant
Masking Description: assigned randomly via ramdom.org
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Application Group (Experimental): Within the scope of the mobile application, information modules on cervical cancer screening tests, cervical cancer risk factors, ways to prevent cervical cancer, types of HPV, and HPV vaccine will be provided. A parallel-group pretest-posttest randomized controlled trial design will be used in the second stage of the study.
  Interventions: Behavioral: Mobile application
- Control Group (No Intervention): The relevant brochures of the Ministry of Health on the prevention of cervical cancer will be given to the experimental and control groups.

INTERVENTIONS:
Behavioral: Mobile application — The mobile application will be designed as a health assistant for women aged between 30-65 to encourage healthy choices and positively develop their behaviors regarding the prevention of cancer. Within the scope of the mobile application, information modules on cervical cancer screening tests, cervical cancer risk factors, ways to prevent cervical cancer, types of HPV, and HPV vaccine will be provided. A parallel-group pretest-posttest randomized controlled trial design will be used in the second stage of the study
  Arms: Mobile Application Group

SUMMARY:
Cervical cancer is one of the most common cancer types affecting women in our country and in the world and causing morbidity. However, the availability of a vaccine for cervical cancer, preventable risk factors and early diagnosis tests offer a unique opportunity to reduce the rate of cervical cancer. In this context, there are studies showing that the practices developed by policies differ and that the classical health approach is insufficient. The effectiveness of the trainings given may vary according to time, place, trainer and personal characteristics of the individual. At the same time, in order to improve the attitudes and behaviours of individuals in terms of prevention and early diagnosis of cervical cancer, awareness of individuals about cervical cancer should be increased. In this way, women will have a say about their own health and their conscious participation in health care services will be realised. Therefore, the aim of this project is to apply cervical cancer awareness training to women and to examine its effect on women's cervical cancer prevention and early diagnosis behaviours. Original value; The fact that there is no mobile application developed for cervical cancer in Turkey reveals the national value of the research. In addition, the mobile application has international unique value as it is the first mobile application structured to provide awareness on cervical cancer prevention and early diagnosis behaviours. The project method was planned for the development and implementation of the mobile application programme. The research design will be a randomised controlled study. The 120 women who meet the inclusion criteria and who apply to more than one family health centre will be randomly assigned to the intervention and control groups. The effect of the mobile application programme on women's attitudes and behaviours towards cervical cancer prevention and early diagnosis will be evaluated at the 6th and 12th weeks. In the evaluation of the data, t-test for independent groups, anova and chi-square tests will be used to measure the effect of the intervention. Widespread effect; In this way, it is planned to reduce the time spent by professionals for care-related activities, to strengthen time management, to provide advantages and improvements in the performance of nurses in patient care management by using technological resources in the health care provided.

DETAILED DESCRIPTION:
Cervical cancer is one of the most common cancer types affecting women in our country and in the world and causing morbidity. However, the availability of a vaccine for cervical cancer, preventable risk factors and early diagnosis tests offer a unique opportunity to reduce the rate of cervical cancer. The World Health Organization launched the "global strategy to accelerate the elimination of cervical cancer as a public health problem" programme in 2020 to eliminate cervical cancer by 2030. In this context, there are studies showing that the practices developed by policies differ and that the classical health approach is insufficient. The effectiveness of the trainings given may vary according to time, place, trainer and personal characteristics of the individual. At the same time, in order to improve the attitudes and behaviours of individuals in terms of prevention and early diagnosis of cervical cancer, awareness of individuals about cervical cancer should be increased. In this way, women will have a say about their own health and their conscious participation in health care services will be realised. Therefore, the aim of this project is to apply cervical cancer awareness training to women and to examine its effect on women's cervical cancer prevention and early diagnosis behaviours. Original value; the fact that there is no mobile application developed for cervical cancer in our country reveals the national value of the research. In addition, the mobile application has an international unique value as it is the first mobile application structured to provide awareness about cervical cancer prevention and early diagnosis behaviours. It is thought that the mobile application programme to be developed has a unique content that provides knowledge and skills to increase the health culture and participation in health decisions thanks to its educational content such as cervical cancer risk factors, prevention methods, diagnostic tests, test results, treatment methods. In addition, it is the first mobile application developed in the national/international field regarding cervical cancer prevention and early diagnosis attitudes and behaviours in line with the deficiencies identified in the literature. The project method was planned for the development and implementation of the mobile application programme. The research design will be a randomised controlled study. A total of 120 women who meet the inclusion criteria and apply to more than one family health centre will be randomly assigned to the intervention (women who use the mobile application programme) and control groups (women who receive the standard education booklet). The mobile application programme includes a total of 12 interfaces for cervical cancer prevention and early diagnosis of cervical cancer. The content of the interfaces and the developed mobile application will be evaluated with the opinion of experts and pre-application. The effect of the mobile application programme on women's attitudes and behaviours towards cervical cancer prevention and early diagnosis will be evaluated in the 6th and 12th weeks. In the evaluation of the data, t-test, anova and chi-square tests for independent groups will be used to measure the effect of the intervention. Widespread effect; In this way, it is planned to reduce the time spent by professionals for care-related activities, to strengthen time management, to provide advantages and improvements in the performance of nurses in patient care management by using technological resources in the health care provided.

ELIGIBILITY:
Inclusion Criteria:

* She applied to Yıldırım Beyazıt Family Health Center and Zafertepe Family Health Center in Kütahya.

  * No pregnancy or malignancy,
  * No hearing and vision problems,
  * Between the ages of 30-65,
  * Having a smart phone,
  * sexually active
  * Can read and write Turkish,
  * Have not had a pap-smear test in the last 5 years,

Exclusion Criteria:

Pregnancy women Breastfeeding Have a history of cancer Have undergone hysterectomy operation Those who have undergone an operation for cervical cancer (cryosurgery, etc.)

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since cervical cancer is seen in women, the study was based on gender.
Enrollment: 120 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Mobile application development | 3 months
  The effectiveness of the mobile application created for cervical cancer awareness will be evaluated with the Mobile Application Usability Scale-MAUS Scale (Mobile Application Usability Scale-MAUS Scale at Week 12). It has a total of 40 items and 7-point Likert type (1=strongly disagree, 7=completely agree). The range of points that can be obtained from the scale is 42-294. The increase in the score indicates that the usability level of the mobile application is high. There are no items that need to be reverse coded in the scale.

SECONDARY OUTCOMES:
effect of the developed mobile application on cervical cancerearly diagnosis attitudes measured by the Attitude Towards Early Diagnosis of Cervical Cancer Scale | 3 months
  The difference between the attitudes towards early diagnosis of cervical cancer of women who use and do not use the mobile application created for cervical cancer awareness will be compared with the mean scores with the Attitude Towards Early Diagnosis of Cervical Cancer Scale. The scale consists of 30 items and is a Likert-type scale. Of the 30 items in the scale, 22 are positive and 8 are negative statements. The scoring of negative statements is reversed. The highest score to be obtained from the scale is 150 and the lowest score is 30.
effect of the developed mobile application on cervical cancer prevention attitudes measured by the Attitude Scale for Cervical Cancer Prevention | 3 months
  Attitude Scale for Cervical Cancer Prevention: consists of 23 items and three sub-dimensions. The items in the scale using Likert-type. The highest score to be obtained from the scale is 115 and the lowest score is 23. The high score obtained from the scale indicates that the individual has high attitudes towards the prevention of cervical cancer
ffect of the developed mobile application on cervical cancer awareness behaviors measured by the Cervical cancer awareness behaviour questionnaire | 3 month
  Cervical cancer awareness behaviors of women using mobile applications will be measured with- Cervical cancer awareness behaviour questionnaire- an 18-question survey prepared by the researcher in line with the literature. Internal consistency tests for the survey were conducted and the Cronbach alpha value was found to be 0.88-0.98.

CONTACTS AND LOCATIONS:
Overall Officials: Sena F Karakışla, MSc, Study Chair — Akdeniz University
Locations (1):
- Kutahya Health Science University, Kütahya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No